CLINICAL TRIAL: NCT06420570
Title: Dysaesthesia Associated With Thoracic Surgery
Brief Title: Sensory Changes Associated With Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC21136
Record Dates: First submitted 2021-11-16; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Surgery
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracic Surgery — Patients will either undergo thoracic surgery, specifically thoracotomy (traditional method of chest surgery using a large surgical incision) or video-assisted thoracic surgery (minimally invasive method using video cameras)

SUMMARY:
Many patients experience chronic pain after thoracic surgery and this is caused by nerve damage during surgery. Changes in skin sensation (dysaesthesia) is typically associated with chronic nerve pain.

We hypothesise that thoracic surgery causes sensory changes. Another hypothesis is that minimally invasive thoracic surgery using video cameras results in less nerve damage and so a smaller area of altered skin sensation, when compared to the traditional method of chest surgery using a large surgical incision. A final hypothesis is that the extent of nerve damage during surgery is associated with the severity of pain early after surgery.

This study is designed to compare the total areas of sensory changes after thoracic surgery on the operated side of the chest with that on the non-operated side of the chest. We also aim to identify the type, pattern, location and area of sensory changes associated with thoracic surgery, comparing the operated with the non-operated side of the chest. In addition, we aim to compare the total area of sensory changes between the traditional method of chest surgery and the minimally invasive method of chest surgery. We would also like to determine whether the severity of pain early after surgery is associated with the area of sensory changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older admitted for elective thoracic surgery

Exclusion Criteria:

* Emergency thoracic surgery
* Thoracic surgery involving sternotomy
* Damage to the spinal cord and/ or intercostal nerves prior to surgery
* Neurological diseases that may alter the skin sensation to the chest wall such as multiple sclerosis and neuropathies, previous surgery of chest wall, a history of chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the thoracic surgery operative list at the Royal Infirmary of Edinburgh.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Area of dysaesthesia on a patient's chest wall | Days after thoracic surgery (at least 3 hours after chest drain removal)
  Areas of dysaesthesia will be detected by applying von frey hair and a sterile, manually blunted 20g hypodermic needle on the patient's chest and back whilst asking the patient to report any sensory changes.
  The areas of dysaesthesia will be marked on chest using different coloured pens for different types of dysaesthesia. The non-operated side of the chest will act as a control. Tracing paper of known weight per unit area will be cut to the same size and shape as the areas of dysaesthesia. Areas of dysaesthesia will be estimated after placing the tracing paper on a sensitive weight scale.

SECONDARY OUTCOMES:
Acute post-operative pain experienced by the patient | Days after thoracic surgery (at least 3 hours after chest drain removal)
  This will be measured using a verbal rating scale: no pain, 0; mild pain, 1; moderate pain, 2; severe pain, 3.

OTHER OUTCOMES:
The patient's mood | Days after thoracic surgery (at least 3 hours after chest drain removal)
  This will be assessed by asking the patient to complete a hospital anxiety and depression questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: R Peter Alston, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared if contacted by email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after completion of study.